CLINICAL TRIAL: NCT01753479
Title: Duodenal Spectroscopy Study for Cancer Diagnosis
Brief Title: Spectroscopy From Duodenum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olympus Corporation (Industry)
Collaborators: M.D. Anderson Cancer Center (Other); Catholic University of the Sacred Heart (Other); Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OMSC-Mag-1
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Test subject (Experimental)
  Interventions: Other: Spectroscopy device

INTERVENTIONS:
Other: Spectroscopy device — Spectrum data are collected using spectroscopy device via an instrumental channel of endoscope. Then spectrum data is analyzed. Numerical features (spectral slope and width of spectrum) are used for statistical analysis.

SUMMARY:
Purpose of this study is to understand the clinical feasibility of duodenal spectroscopy to adenocarcinoma patients.

DETAILED DESCRIPTION:
Pancreatic cancer (PC) is the most lethal of all major cancers with a five year survival rate of 5 %. While stage I and II tumors leads to an improvement in survival, almost all PCs are currently diagnosed at more advanced non-resectable stages since minimally invasive technique which is capable of screening early-stage PC does not exist. Serum CA19-9 is not recommended as a screening technique because of its low sensitivity and specificity. Imaging modalities such as MRI, CT, EUS and ERCP are more accurate but are not appropriate screening tools due to their high cost, discomfort and complications. Therefore, there is a strong demand for a screening tool with high sensitivity and specificity which is highly acceptable for the patient. The investigators would like to look at the spectroscopy technique for pancreatic cancer diagnosis via an upper endoscopy. A definite diagnosis of the patient is made with histology, cytology or imaging diagnosis. Therefore this study can be positioned as a feasibility study.

ELIGIBILITY:
Inclusion Criteria:

* Common inclusion criterion

  * Age is 18 years or older.
  * Informed consent was obtained.
  * Inclusion criterion for normal cohort
  * An upper GI endoscopy is scheduled to check upper abdominal symptoms.
  * No findings of pancreatic disorder as documented by CT or MRI or EUS
* Inclusion criterion for PC suspicious cohort * A EUS or ERCP is scheduled to suspected pancreatic disorder.

Exclusion Criteria:

* Common exclusion criterion

  * Severe cardiac disease
  * Severe respiratory disease
  * Bleeding disorders
  * Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
The spectral data of the normal cohort and UICC stage II pancreatic ductal adenocarcinoma cohort | 1 year
  To clarify that there is the statistically-significant difference between two cohorts.

SECONDARY OUTCOMES:
The sensitivity and specificity to detect UICC stage II pancreatic ductal adenocarcinoma among all participants. | 1 year
  A receiver operating characteristic (ROC) is evaluated. A cut-off is then chosen from this ROC curve to maximize both sensitivity and specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Wallace, M.D., Principal Investigator — Mayo Clinic
Locations (4):
- United States (2):
  - Mayo Clinic Florida, Jacksonville, Florida
  - The University of Texas M. D. Anderson Cancer Center, Houston, Texas
- Hôpital Erasme, Brussels, Brussels Capital, Belgium
- Università Cattolica del Sacro Cuore, Rome, Lazio, Italy